CLINICAL TRIAL: NCT03836079
Title: Superior Vena Caval Occlusion in Subjects With Acute Decompensated Heart Failure
Brief Title: SVC Occlusion in Subjects With Acute Decompensated Heart Failure
Acronym: VENUS-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 101773-002
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Acute Decompensated Heart Failure; Acute Heart Failure; Congestive Heart Failure; Heart Diseases
MeSH Terms: conditions — Heart Failure; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- ADHF Patients (Experimental): Treatment with preCARDIA System
  Interventions: Device: preCARDIA system

INTERVENTIONS:
Device: preCARDIA system — Intermittent occlusion of the SVC

SUMMARY:
Safety and performance evaluation of the preCARDIA System for patients with ADHF.

DETAILED DESCRIPTION:
The objective of this early feasibility study is to evaluate the safety and performance of the preCARDIA System for Superior Vena Caval (SVC) intermittent mechanical occlusion as a therapeutic approach in significantly congested subjects with Acute Decompensated Heart Failure (ADHF), who are not diuresing adequately.

ELIGIBILITY:
Inclusion Criteria:

* NYHA Class III-IV heart failure
* Subjects with inadequate diuresis
* Stage C-D systolic heart failure

Exclusion Criteria:

* Active myocardial ischemia or acute coronary syndrome (ACS)
* Severe aortic or mitral valve insufficiency
* Severe peripheral vascular disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Freedom from Major Adverse Events through 90 days post-discharge. | 90 days post-discharge
  MAE is defined as death, myocardial infarction, major thromboembolic event, vascular damage requiring surgical intervention, hemorrhagic stroke or prolongation of heart failure- related hospitalization attributable to the preCARDIA device or procedure.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Colorado Heart & Vascular, Lakewood, Colorado
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Tampa General Hospital, Tampa, Florida
  - Northwestern, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Kansas University Medical Center, Kansas City, Kansas
  - Tufts Medical Center, Boston, Massachusetts
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - CentraCare Heart & Vascular Center, Saint Cloud, Minnesota
  - OhioHealth, Columbus, Ohio
  - Providence Health & Services, Portland, Oregon
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist, Houston, Texas
  - Baylor, Scott & White Medical Center - Temple, Temple, Texas
  - Inova Health System, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kapur NK, Kiernan MS, Gorgoshvili I, Yousefzai R, Vorovich EE, Tedford RJ, Sauer AJ, Abraham J, Resor CD, Kimmelstiel CD, Benzuly KH, Steinberg DH, Messer J, Burkhoff D, Karas RH. Intermittent Occlusion of the Superior Vena Cava to Improve Hemodynamics in Patients With Acutely Decompensated Heart Failure: The VENUS-HF Early Feasibility Study. Circ Heart Fail. 2022 Feb;15(2):e008934. doi: 10.1161/CIRCHEARTFAILURE.121.008934. Epub 2022 Jan 10. PMID 35000420